CLINICAL TRIAL: NCT04085796
Title: An Exploration of the Lived Experience of Receiving and Providing an Intentional Compassionate Communication Intervention (ICCI) for Older People While in Accident and Emergency Department
Brief Title: ICCI for Older Patients in A&E
Status: Completed | Type: Observational
Sponsor: Bournemouth University (Other)
Responsible Party: Principal Investigator, Marta Paglioni, Dramatherapist, PhD student, Bournemouth University
Other Study IDs: 22232
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Older Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older patients: Older patients who received the ICCI while in the hospital's A&E
  Interventions: Other: ICCI
- ICCI Professional: The member of staff who delivers the ICCI at the site
  Interventions: Other: ICCI

INTERVENTIONS:
Other: ICCI — Intentional Compassionate Communication Intervention

SUMMARY:
Study Objectives

1. To gather rich, evocative accounts of older patients aged 65 years and over -who may have felt disorientated in the Accident and Emergency department (A&E) of a district hospital and who received an Intentional Compassionate Communication Intervention (ICCI)- about their personal experience of the A&E
2. To gather rich and evocative accounts of a member of staff who delivers an Intentional Compassionate Communication Intervention (ICCI) to older people in the A&E of a district hospital about their personal experience of doing so.

DETAILED DESCRIPTION:
1.1 Background The number of hospital emergency admissions has dramatically increased in England, by 42%, over the last 12 years (The Health Foundation 2018). Qualitative research published between 1990 and 2006 on the patient experience within the emergency department showed that most patients arrived at the A&E with the perception that their injury or condition was serious or life threatening (Baraff et al. 1992; Olsson and Hansagi 2001; Nystrom et al. 2003) and this perception was often accompanied by physical pain (Britten and Shaw 1994). The situation is one in which patients feel vulnerable, anxious, stressed and fearful (Olsson and Hansagi 2001; Kihlgren et al. 2004).

In the UK, nearly a quarter of the people arriving at A&E are over 65 years (Geddes 2013), older patients represent a demographic group whose emergency admissions have seen a particularly sharp rise over the last 12 years, especially patients aged 85 years or older (The Health Foundation 2018). This entails hospital staff having to deal in the emergency situation with patients presenting with much more complex needs associated with co-morbidities and often with less external support than younger people (Sorrel 2010).

Older patients are more prone to feel disorientated in A&E. This can be due to a high percentage of them presenting with dementia, delirium, delirium superimposed on dementia or other CSD (Cognitive Spectrum Disorders), and they are also at higher risk of developing delirium while in the emergency department (Reynish et al. 2017). Delirium is a common medical problem that is characterised by changes in cognitive function. When delirium occurs, people are confused. Its onset is quite sudden, but it usually lasts only for a few days (NHS 2018). However, if not addressed delirium can become a serious complication which can lead to longer length of stay in hospital and higher mortality (Witlox et al. 2010). Stress is one of the common triggers for delirium and there is also some evidence that longer and particularly stressful A&E experiences are associated with the risk of older patients developing delirium over the following hours (Bo et al. 2016).

There have been a few published studies exploring the experiences of A&E from the specific point of view of older patients which report that most of them believe that their symptoms pose a serious threat to their life or to the control they exert over their lives (Olsson and Hansagi 2001; Kihlgrenet al. 2004) and that the attitudes of nurses in A&E are often perceived as indifferent and inattentive, thus causing a feeling of exclusion and disappointment (Olofson et al. 2012). Empathy and compassion are perceived by patients to be the most significant elements of good care in A&E (Kihlgren et al. 2005).

Compassionate Care is not a new concern for the NHS but following high profile failings (Francis 2013) government policies such as the Compassionate Care in the NHS (Department of Health 2015) have been introduced, further emphasising the importance of humanised care (Todres et al. 2009). Recent literature has explored different perspectives, from the poor experiences of care by older people living with frailty which, has been uncovered by the Francis Report (Singh et al. 2013), to the challenges experienced by nurses expected to deliver compassionate care, who often struggle to align the reality of practice to their ideals (Curtis et al. 2012).

Cornwell and Goodrich (2009 p.15), in a study exploring patients' experiences state: "the presence or absence of compassion often marks the lasting and vivid memories patients and family members retain about the overall experience of care in hospital". This is valid also for patients who are temporarily confused and/or live with dementia. Projects like the "Dementia diaries" project, show that people can not only be aware of how they are treated and how they feel even in the middle of an extremely confused state, but they can also be able to recall this (Agnes' story 2018). Patient satisfaction should be considered a goal in itself; however, the literature also suggests that patients receiving clear and compassionate communication are more likely to disclose their symptoms enabling greater understanding of their situation and more accurate diagnoses (Epstein et al. 2005 and Cornwell and Goodrich 2009).

The evidence from the paragraphs above indicates that an investment in targeted compassionate communication for older people in A&E could make their care more effective, with the potential to reduce complications and make healthcare delivery more economically sustainable for the NHS alongside giving patients and their families a better experience.

The awareness of the high incidence of stress in A&E, and of the importance of compassionate care for older people has driven the development of a specific Intentional Compassionate Communication Intervention (ICCI) within the A&E of a district hospital. The ICCI comprises proactive communication-focused support to older people. It involves a member of staff taking responsibility for the ICCI to meet older patients' psychological needs and relieve their anxieties through talking to them, sharing information with them and reassuring them when in A&E.

The delivery of the intervention gives priority to support older people who are in A&E alone and to those of them who appear to be cognitively impaired. The aim is to provide patients who may feel disorientated additional support in order to reduce the anxiety associated with being in A&E. Using effective communication skills the member of staff demonstrates compassion and empathy to the older patients whilst they are in a busy A&E department. Activities may include talking to them, gently re-orientating them if confused, by asking simple questions while using a friendly and reassuring tone of voice, offering a glass of water or a cup of tea, maybe a blanket. The member of staff can also try to reassure patients by enquiring with other staff about the outcome of an examination or about the next step into the patient's hospital stay when it happens to be too busy or staff is under too much pressure to be able to communicate with patients promptly and efficiently.

She also holds many hands, because of pain or because of fear. She purposefully uses a sense of humor to prompt a smile or a quick laugh. If words are not helpful (because the cognitive impairment is too severe, for example) she might play some music using an I-pad or bringing some soft toys for patients to cuddle. What lays at the basis of this intervention is the meeting between two human beings whereas one of them is in pain (psychological and often also physical) and the other one somehow "feels" that pain and has a genuine wish to relieve it. The ICCI is totally person-centered and does not rely on any particular technique, rather it is exclusively based on a shared, deeply human drive.

A systematic review of literature Sonis et al. 2017) highlighted that most recent studies of patient experiences at A&E are quantitative and use methods such as surveys or interviews, concentrating on judgments of patients after their A&E visit. A few qualitative studies have been carried out. Baraff et al. (1992) showed that patients are very concerned about losing autonomy and independence, and Olthuis et al. (2014) showed that during the A&E stay patients not only have to deal with their disorder, its consequences, and the situation they are in, but they are also continuously troubled by all kinds of matters. They found that it is a struggle for them to admit that something is wrong with them, to trust the health care professionals, to endure waiting periods, to have a blood sample taken, to undress, to deal with their relatives and reassure them, and even to get something to drink or eat.

Despite this, we still do not know very much about disorientated patients experiences in A&E. Considering the above, and that there are few studies focusing on the lived experience of older patients in A&E but currently no published studies that focus on the experience of Intentional Compassionate Care Interventions (ICCI) within A&E, improved understanding of the lived experience of patients with regards to the provision of ICCI within A&E would be of great value in nursing; particularly considering that the experience of older people in A&E is often characterized by discomfort, fear, and pain, and can trigger disorientation and confusion. Moreover, people with Dementia or other cognitive impairments have a unique contribution to make in research. Hearing their voices can help people see the A&E experience from their point of view, contributing to fight the assumptions and the stigma often associated with such a diagnosis (Alzheimer's Society 2018).

1.2 Clinical Data In the UK, nearly a quarter of the people arriving at A&E are over 65 years (Geddes 2013) and older patients represent a demographic group whose emergency admissions have seen a particularly sharp rise over the last 12 years (The Health Foundation 2018). The experience of older people in the A&E is often characterised by discomfort and anxiety (Baraff et al. 1992; Olsson and Hansagi 2001; Kihlgrenet al. 2004; Olofson et al. 2012). Stressful experiences may represent a possible trigger for delirium, a common and significant complication between older hospital patients which can affect the following course of recovery and the overall hospital length of stay (Cunningham and MacLullich 2013). There is some evidence that longer and particularly stressful A&E experiences are associated with the risk of older patients developing delirium over the following hours (Bo et al. 2016).

Compassionate care seems to reduce patient anxiety (Gilbert and Procter 2006 and studies conducted in A&E show that empathy and compassion are the most significant elements of good care for older patients in A&E (Kihlgren et al. 2005).

1.3 Rationale

The results of the research will contribute to a deeper understanding of older potentially disoriented patients' lived experiences of being in A&E and receiving an A&E based ICCI. This study could impact upon NHS consideration of possible new roles in A&E that are responsible for ICCI and how to make older patients' care more effective and sustainable, and give this patient group a better experience and outcome. Including people living with dementia or experiencing other cognitive disorders in the study is not only a way to improve their care, but also a way of valuing their contribution to society.

1.4 Risks/Benefits During the study patient participants will have the opportunity to reflect on their experience of being in A&E, on their emotional needs and if and how these were met during their period in A&E. Reflecting and acknowledging our need for human connection and meaningful interactions raises our awareness and this can translate into a benefit for these participants.

The recruitment of patient participants for interview may include those living with dementia or other cognitive impairments and it is recognised that they represent a vulnerable population. However, only those who have been identified as being able to give informed consent by a registered health care professional member of the Dementia Care Team, will be invited to participate to the study.

The researcher will remain sensitive to any sign of distress during the interview and suspend or stop their participation if indicated. Taking extra-care when interacting with vulnerable people is essential, however, excluding patients living with dementia from participation in research interviews could represent a form of discrimination, as their voice would seldom be heard in research and by the services they use. Lack of capacity can make people with dementia particularly vulnerable to discrimination (Alzheimer's Society 2018) and this is also valid for their participation to research. Under the Mental Capacity Act a person is presumed to be able to make their own decisions "unless all practical steps to help them to make a decision have been taken without success" (Mental Capacity Act 2005).

When interacting with another person like during an interview, there is always a degree of risk of exposure to the Covid19 virus or other viruses for both the participant and the researcher. However, to minimise the risk for both parts, the researcher will only approach participants who have already been tested negative for Covid19 at their admission to the ward, and will do so in a Covid-Cold ward (where only patients tested negative to Covid19 are admitted, and where patients are regularly tested for Covid19.). She will approach them only after having carefully washed her hands and while wearing the appropriate PPE in place at the hospital. She will also maintain the appropriate safety distance suggested by the latest UK Government guidelines, and will not have any physical contact with the participant. The interview will last a maximum of 40 minutes to minimise the risk.

The researcher will not travel to the hospital if she develops symptoms of Covid19.

Also, the professional delivering the ICCI will be asked to participate in a series of online interviews about their experience (it is expected to run around 3 to 5 interviews which are expected to take place weekly) using a secure online platform, assessed and chosen following GDPR principles, and the same criteria of informed consent and freedom to withdrawn will apply too. The questions might touch on sensitive issues for the professional, and the researcher will remain sensitive to any sign of distress during the interview and suspend or stop their participation if indicated, also offering them emotional support. If further support is needed, she will signpost them to appropriate psychological support services.

The researcher will use good practices to ensure maximal security: the researcher will make sure to connect via a BU laptop which has all the required firewalls in place and that their internet connection is protected and will ask the professional to ensure her connection is similarly protected. the researcher will make sure that the online platform used for the online meeting is secure enough following GDPR principles and she will personally password protect and lock each meeting as soon as it starts. She will make sure that nobody else is in the room with her and will ask the ICCI professional to do the same to protect confidentiality. In addition, the researcher will make use of headphones so that there is no chance of participant being overheard, and will advise the participant to do the same.

2. Study Objectives and Design 2.1 Study Objectives

1. To gather rich, evocative accounts of older patients aged 65 years and over -who may have felt disorientated in the Accident and Emergency department (A&E) of a district hospital and who received an Intentional Compassionate Communication Intervention (ICCI)- about their personal experience of the A&E;
2. To gather rich and evocative accounts of a member of staff who delivers an Intentional Compassionate Communication Intervention (ICCI) to older people in the A&E of a district hospital about their personal experience of doing so.

2.2 Study Endpoint The end point will be the completion of the qualitative analysis of transcripts from patients' interviews and the ICCI professional's interviews, when enough rich data to answer the research questions have been collected.

2.3 Study Design This is a qualitative study whose aim is to explore the lived experience of a sample of older patients (65 years and over) who may have felt disoriented in the A&E of a district hospital and who received an ICCI.

Using Interpretative Phenomenological Analysis (IPA), in-depth interviews will be carried out with up to 15 patients and the professional delivering the ICCI at the site, and the data created from the transcripts will be analysed thematically.

2.4 Recruitment and consent: The researcher has spent more than one year collaborating with the Dementia Care Team both providing emotional support to patients at bedside and supporting staff and volunteers in relating to older patients in hospital. She also ran informal observations of the ICCI delivered in A&E to orientate herself to the setting. As a result of this she developed a network of gatekeepers and has access to the wards and to different professionals, particularly in the context of the Dementia Care Team.

The Dementia Care Team will identify possible participants for the study across different wards in the hospital. An appropriately qualified professional member of the Dementia Care Team will assess participant's mental capacity specifically around the decision to consent to participate to the research at all three key points in the study: a) at introduction b) immediately before Informed Consent is given and c) immediately before the interview.

At introduction, after patients' permission for the researcher to visit them has been gained by a member of the care team, the researcher will approach them to give oral and written information (Participant Information Sheet V.6) and to ask for consent. This will happen in a so called Cold-Covid ward (where only patients tested negative for Covid19 are admitted) only when the care team has considered them physically and mentally fit for this and they have been tested negative for Covid19. In accordance with the Mental Capacity Act, the professional will verify if the patient is able to understand, retain, use and weight the information provided and to communicate his decision (Mental Capacity Act 2005).

Patients will be given as much time as they need to make their decision on whether to participate.

The professional delivering the ICCI will be initially approached by email -to their secure NHS trust email address- by the researcher's clinical supervisor to ask if they want to consider participate. If they agree, they will be given the researcher's contact details. When the professional will have contacted the researcher, they will be given all information needed about the study and their participation. If they still want to go ahead, they will receive a copy of a specific PIS (Participant Information Sheet for ICCI Professional V.1) and they will be allowed to ask any question via telephone or email and as much time as they need to make their decision. If they decide to participate, hey will then receive a copy of a specific ICF (ICF for ICCI professional V.1) and only after they will have signed it -in accordance with HRA and MHRA joint statement on seeking consent by electronic methods 2018 a typed electronic signature is sufficient for this study- and send it back to the researcher, an appointment for the first interview will be booked.

It is recognized that there is the potential for feelings of coercion in the workplace when asking a member of staff to take part to a study like this. With this in mind, it will be made very clear -both verbally and in the PIS- to the person involved, that there is no obligation for them to participate, and that if they refuses, that will not have any impact on them, on their job, or on their relationships with their manager and colleagues.

ELIGIBILITY:
Inclusion criteria For Patients:

* Patients aged 65 years and over;
* Admitted for any reason to the hospital via A&E;
* Patients presenting either alone or confused or with a diagnosis of dementia;
* Patients who received the ICCI while in A&E;
* Patients referred to the Dementia Care Team (which support patients admitted into the hospital who have a cognitive impairment either as a result of an underlying dementia -diagnosed or otherwise- or who are experiencing transitory cognitive symptoms such as confusion as a result of a delirium);
* Patients who are able to give informed consent to participate in the study as identified by a registered health care professional
* Patients who have been tested for Covid19 at admission to the ward and who are in a Cold-Covid ward

Inclusion criteria for the member of staff:

-The professional who has delivered the ICCI at the site over the last 3 years.

Exclusion criteria For Patients:

* Patients who cannot give informed consent;
* Patients with a physical condition that is immediately life-threatening or unstable;
* Patients involved in other clinical trials which present a significant burden to them.
* Patients who tested positive for Covid19

Exclusion criteria For the member of staff:

-If the member of staff is unable or unwilling to participate for any reason.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Older patients who present to the the A&E alone, or confused, or with a diagnosis of Dementia and who receive an ICCI when in A&E;
  The Professional who has been delivering the ICCI to older people in A&E over the past 4 years.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
The lived experience of older people receiving an ICCI while in A&EI people A&E | 1 year
  personal lived experience ( this is a qualitative study)
The lived experience of the professional delivering the ICCI to older people in A&E | 4 months
  personal lived experience ( this is a qualitative study)

CONTACTS AND LOCATIONS:
Locations (1):
- South West NHS Trust, Bournemouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No